CLINICAL TRIAL: NCT03548649
Title: Clinical Research for Exoskeleton Robot
Brief Title: The Efficacy and Safety of a New Power Exoskeleton Robot for Improving Walking Ability in Spinal Cord Injury Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: The Industrial Technology Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-03-012C
Record Dates: First submitted 2017-08-05; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Spinal Cord Injuries; Complete Spinal Cord Injury; Incomplete Spinal Cord Injury
Keywords: spinal cord injury; complete spinal cord injury; incomplete spinal cord injury; exoskeleton robot; gait training; security testing; functional testing
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: AIS A-D SCI patients with injury level C7-L5
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exoskeleton robot training group (Experimental): subjects will receive exoskeleton robot training for 20 sessions (1 hr/session).
  Interventions: Device: exoskeleton robot training

INTERVENTIONS:
Device: exoskeleton robot training — subjects will learn to independently use the exoskeleton robot to perform functional activities (including stand-up, sit-down, stepping forward, and walking).
  Other Names: gait training

SUMMARY:
In Taiwan, there are more than 23,000 individuals with spinal cord injuries (SCI, mean age: 27 years), with an increment of new 1,200 SCI individuals each year. Recovery of ambulatory function is among the most important therapeutic goals because 92% of the individuals with SCI have to use the wheelchair for the rest of their lives.

The lower limb powered exoskeleton robot, FREE Walk, used for training in this research was developed by FREE Bionics Inc. The main purpose of this research is to test the safety and feasibility of FREE Walk exoskeleton robot. In addition, the research will further investigate the range of injury levels for the intended SCI users and the learning time needed for the users to independently operate the exoskeleton robot.

DETAILED DESCRIPTION:
Individuals with SCI who meet the inclusion criteria will be referred to the investigators. Participants will be given consent forms and explained the research before participating. The participants must pass the initial evaluation described below in order to go through robot training: (1) medical history, (2) bone density, (3) joint range of motion, ROM (4) strength (manual muscle test, MMT), (5) muscle tone (modified Ashworth scale, MAS).

The training program consists of 5-min preparation, 50-min of functional activities training including weight shifting, sit-down, stand-up, stepping and walking, and 5-min training feedback. Every participant will receive at least 20 training sessions (1 hour per session, 2-5 sessions per week) and an post-training evaluation after completion of training. The post-training evaluation includes the following tests: timed up-and-go test, 10-meter walk test, and 6-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

1. Spinal cord injury patients whose injury levels range from C7 to L5, ASIA impairment scale A to D, can use forearm crutch and can't walk without an assistive device.
2. In a stable condition, for example, at least 3 months after first injury/onset, or with stable spine, or had been corrected (internal fixation).
3. Age between 18-70.
4. height between 150-190cm; weight less than 100kg; thigh length between 32-47cm; leg length (from lateral epicondyle of femur to sole) between 23-59cm.
5. Normal joint range of motion(ROM) of both lower extremities and upper extremities or ROM limitation will not affect ambulation.
6. Can maintain trunk stability with or without hand support in sitting position for 60s.

Exclusion Criteria:

1. Combine other neurological diseases, for example, stroke, cerebral palsy, Parkinson's disease,... etc.
2. Femoral T-score <-2.5. (Doctor's approval must be obtained for those who with femoral t-score between -2.5 and -3).
3. Other medical conditions which will affect weight bearing or ambulation.
4. Medical history including fracture(due to osteoporosis in the past 2 years), heart failure, myocardial infarction.
5. Skin conditions including allergy, pressure sore, infection, ...etc.
6. Impaired mental or cognitive conditions that will affect training or evaluation.
7. Severe contracture or limited joint range of motion of lower extremities.
8. Severe spasticity which will impede the movement of exoskeleton robot.
9. Heterotopic ossification.
10. non-union fracture or open wound.
11. pregnancy.
12. other conditions that is not applicable for use the exoskeleton robot.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
10 meters walking test | Test will be held before starting the first training session and after completing 20 training sessions.(1 hour per session)
  Subjects walk with exoskeleton for 10 metres, with the time measured for the intermediate 6 metres to allow for acceleration and deceleration.

SECONDARY OUTCOMES:
timed up-and-go test | Test will be held before starting the first training session and after completing 20 training sessions.(1 hour per session)
  Record the time needed to perform timed up-and-go test wearing exoskeleton robot
6-minutes walking test | Test will be held before starting the first training session and after completing 20 training sessions.(1 hour per session)
  Record the distance covered to perform 6-min walk test wearing exoskeleton robot. Rate of Perceived Exertion will be recorded at the end of the 6-min walk test to evaluate users' endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-An Tsai, MD, Study Chair — 0938-592-575
Locations (1):
- Taipei Venterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] van Hedel HJ, Wirz M, Dietz V. Assessing walking ability in subjects with spinal cord injury: validity and reliability of 3 walking tests. Arch Phys Med Rehabil. 2005 Feb;86(2):190-6. doi: 10.1016/j.apmr.2004.02.010. PMID 15706542
- [Background] Harada ND, Chiu V, Stewart AL. Mobility-related function in older adults: assessment with a 6-minute walk test. Arch Phys Med Rehabil. 1999 Jul;80(7):837-41. doi: 10.1016/s0003-9993(99)90236-8. PMID 10414771
- See also: World Health Organization — http://www.who.int/mediacentre/factsheets/fs384/en/
- See also: foundation of spinal cord injury, R.O.C — http://www.fsci.org.tw/ap/news_view.aspx?bid=21&sn=6907d6d9-18ec-4901-bca4-aa56065444a9